CLINICAL TRIAL: NCT01448850
Title: A Phase 2 Double-blind, Placebo-controlled Study to Evaluate the Efficacy of MEDI8968 in Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Efficacy of MEDI8968 in Chronic Obstructive Pulmonary Disease
Acronym: SPRING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CD-RI-MEDI8968-1103
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD); MEDI8968
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to MEDI8968 as IV infusion on Day 1 followed by SC injection every 4 weeks up to Week 53.
  Interventions: Other: Placebo
- MEDI8968 600 mg IV, 300 mg SC (Experimental): MEDI8968 600 milligram (mg) as intravenous (IV) infusion on Day 1 followed by 300 mg injection subcutaneously (SC) every 4 weeks up to Week 53.
  Interventions: Biological: MEDI8968 600 mg IV, 300 mg SC

INTERVENTIONS:
Biological: MEDI8968 600 mg IV, 300 mg SC — MEDI8968 600 mg as IV infusion on Day 1 followed by 300 mg injection SC every 4 weeks up to Week 53.
  Arms: MEDI8968 600 mg IV, 300 mg SC
Other: Placebo — Placebo matched to MEDI8968 as IV infusion on Day 1 followed by SC injection every 4 weeks up to Week 53.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of MEDI8968 on the rate of moderate or severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD) in adult subjects with symptomatic, moderate to very severe COPD (Global Initiative for Chronic Obstructive Lung Disease - GOLD stage II-IV) receiving standard maintenance therapy for the underlying disease condition.

DETAILED DESCRIPTION:
A Phase 2 double-blind, placebo-controlled study to evaluate the efficacy of MEDI8968 in Chronic Obstructive Pulmonary Disease. The study will have a screening phase of 23 days, treatment phase from Week 1 to 53 and follow-up phase from Week 53 to 69. Participants will receive either MEDI8968 600 milligram (mg) as intravenous (IV) infusion on Day 1 followed by 300 mg injection subcutaneously (SC) every 4 weeks up to Week 53 or matching placebo in the same fashion. Participants will primarily be assessed for incidence rate of moderate or severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD). Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 through 75 years
* Predicted (Global Initiative for Chronic Obstructive Lung Disease [GOLD] stage II, III, and IV) at Screening
* History of previous acute exacerbations of chronic obstructive pulmonary disease (AECOPD) 12 months prior to Screening
* Clinically stable and free from an AECOPD for 8 weeks prior to Day 1
* Current smoker or ex-smoker with a tobacco history of more than or equal to (>=) 10 pack-years.

Exclusion Criteria:

* Past or present disease or disorder,
* Significant or unstable ischemic heart disease etc
* Known history of allergy or reaction to any component of the investigational manufacturing product (IMP)
* Past or current malignancy within the past 5 years
* Subjects have had a chest x-ray or Computed Tomography (CT) scan suggestive of malignancy or tuberculosis (TB).
* Use of immunosuppressive medication receipt of any biologic agent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rene Van Der Merwe, MBChB, MFPM, Study Director — MedImmune Ltd
Locations (60):
- United States (12):
  - Research Site, Peoria, Arizona
  - Research Site, Clearwater, Florida
  - Research Site, Duluth, Georgia
  - Research Site, Auburn, Maine
  - Research Site, Buffalo, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Richmond, Virginia
- Bulgaria (5):
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Veliko Tarnovo
- Czechia (6):
  - Research Site, Brno
  - Research Site, Jindřichův Hradec
  - Research Site, Karlovy Vary
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Strakonice
- Hungary (11):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Farkasgyepü
  - Research Site, Komárom
  - Research Site, Mátészalka
  - Research Site, Mátraháza
  - Research Site, Mosonmagyaróvár
  - Research Site, Nagykanizsa
  - Research Site, Szikszó
  - Research Site, Tatabánya
  - Research Site, Törökbálint
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Quezon City
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Oświęcim
  - Research Site, Poznan
  - Research Site, Wroclaw
  - Research Site, Zgierz
- Ukraine (7):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Simferopol
  - Research Site, Vinnytsia
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Newcastle upon Tyne
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Calverley PMA, Sethi S, Dawson M, Ward CK, Finch DK, Penney M, Newbold P, van der Merwe R. A randomised, placebo-controlled trial of anti-interleukin-1 receptor 1 monoclonal antibody MEDI8968 in chronic obstructive pulmonary disease. Respir Res. 2017 Aug 9;18(1):153. doi: 10.1186/s12931-017-0633-7. PMID 28793896

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 464 participants were screened and 324 participants were randomized into the study.
Groups:
- Placebo: Placebo matched to MEDI8968 as intravenous (IV) infusion on Day 1 followed by subcutaneous (SC) injection every 4 weeks up to Week 53.
- MEDI8968 600 mg IV, 300 mg SC: MEDI8968 600 milligram (mg) as IV infusion on Day 1 followed by 300 mg injection SC every 4 weeks up to Week 53.
Period: Overall Study
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Started | 164 | 160
Completed | 130 | 120
Not Completed | 34 | 40
Not completed — Death | 3 | 6
Not completed — Withdrawal by Subject | 13 | 21
Not completed — Lost to Follow-up | 3 | 1
Not completed — Other | 15 | 12

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all participants who were randomized into the study and received any investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC | Total
Number analyzed (Participants) | 164 | 160 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (6.8) | 62.8 (6.7) | 62.9 (6.8)
Gender [Count of Participants; unit: Participants]
  Female | 54 | 50 | 104
  Male | 110 | 110 | 220

OUTCOME MEASURES:

1. Primary Outcome: Mean Rate of Moderate or Severe Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: An AECOPD is defined as worsening of two or more major symptoms or one major and one minor symptom for two or more consecutive days. The severity of an AECOPD is defined as: Moderate exacerbations require treatment with systemic corticosteroids, and or antibiotics. Severe exacerbations require hospitalization. The AECOPD rate was analyzed using a Poisson Regression model adjusted for over dispersion with number of exacerbations as the outcome and the log of follow-up time as an offset variable, with covariates for treatment group (MEDI8986, placebo), background maintenance therapy and previous exacerbations. Mean exacerbations were presented as number of exacerbations/year.
Time Frame: Day 1 up to 393
Population: as for baseline characteristics
Measure: Mean (90% Confidence Interval); unit: AECOPD events/year
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 164 | 160
AECOPD events/year | 0.78 [0.63 to 0.96] | 0.71 [0.57 to 0.90]
Statistical Analysis 1: Comparison: Placebo vs MEDI8968 600 mg IV, 300 mg SC; Test type: Superiority or Other; p = 0.645, Poisson regression — Data was analyzed using Poisson regression with Pearson correction, adjusting for treatment, background therapy and history of previous exacerbations; Rate ratio = 0.92, 90% CI 2-sided [0.68 to 1.25]

2. Secondary Outcome: Mean Rate of Severe Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: An AECOPD is defined as worsening of two or more major symptoms or one major and one minor symptom for two or more consecutive days. Severe exacerbations require hospitalization. The AECOPD rate was analyzed using a Poisson Regression model adjusted for over dispersion with number of exacerbations as the outcome and the log of follow-up time as an offset variable, with covariates for treatment group (MEDI8986, placebo), background maintenance therapy and previous exacerbations. Mean exacerbations were presented as number of exacerbations/year.
Time Frame: Day 1 up to 393
Population: The mITT population included all participants who were randomized into the study and received any investigational product.
Measure: Mean (90% Confidence Interval); unit: AECOPD events/year
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 164 | 160
AECOPD events/year | 0.14 [0.09 to 0.21] | 0.10 [0.06 to 0.16]

3. Secondary Outcome: Time to First Moderate or Severe Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: Time to first worsening of two or more major symptoms or one major and one minor symptom for two or more consecutive days. The severity of an AECOPD is defined as: Mild exacerbations require treatment with an increase in usual therapy, e.g., increase use of short acting bronchodilators. Moderate exacerbations require treatment with systemic corticosteroids, and or antibiotics. Severe exacerbations require hospitalization.
Time Frame: Day 1 up to 393
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 164 | 160
days | NA [173.0 to NA] — Median and upper limit of 95% confidence interval (CI) were not evaluable as less than 50% of the participants had moderate or severe AECOPD. | NA [134.0 to NA] — Median and upper limit of 95% confidence interval (CI) were not evaluable as less than 50% of the participants had moderate or severe AECOPD.

4. Secondary Outcome: Change From Baseline in COPD-Specific Saint George's Respiratory Questionnaire (SGRQ-C) Total and Subscales Scores at Week 53
Description: The SGRQ is a health related quality of life questionnaire consisting of 40 items in three domains: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Each question's response has a unique empirically derived weight where lowest possible weight is zero and the highest is 100. The total score and domain score are derived from the relevant items and converted to a score of 0 to 100 with a higher score indicating poorer health status.
Time Frame: Baseline and Week 53
Population: The mITT population included all participants who were randomized into the study and received any investigational product. Here, 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 164 | 160
units on scale
  Change at Week 53: Total Score (n=134, 123) | -2.76 (1.069) | -2.22 (1.101)
  Change at Week 53: Activity Score (n=134, 123) | -1.15 (1.306) | -1.38 (1.348)
  Change at Week 53: Impacts Score (n=134, 123) | -2.91 (1.326) | -1.08 (1.366)
  Change at Week 53: Symptoms Score (n=134, 123) | -5.60 (1.279) | -6.81 (1.325)

5. Secondary Outcome: Percentage of Participants With Improvement in COPD-Specific Saint George's Respiratory Questionnaire (SGRQ-C) Total Score
Description: The SGRQ is a health related quality of life questionnaire consisting of 40 items in three domains: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Each question's response has a unique empirically derived weight where lowest possible weight is zero and the highest is 100. The total score and domain score are derived from the relevant items and converted to a score of 0 to 100 with a higher score indicating poorer health status. A 4-point change in total score demonstrates a clinically meaningful change, while an 8-point change and a 12-point change are interpreted as a moderate and large change in health status, respectively.
Time Frame: Week 53
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 164 | 160
percentage of participants
  Week 53: 4-point improvement (n=134,123) | 45.5 | 43.1
  Week 53: 12-point improvement (n=134,123) | 17.9 | 17.1

6. Secondary Outcome: Change From Baseline in Body Mass Index, Airflow Obstruction, Dyspnea, and Exercise Capacity (BODE) Score at Week 53
Description: The BODE index is a multi-dimension COPD grading system that incorporates body-mass index (B), degree of airflow obstruction (O), dyspnea (D), and exercise capacity (E) as measured by the modified medical research council (MMRC) dyspnea scale and the 6-minute walk test. The MMRC dyspnea scale is a 5-point scale that measures the level of dyspnea (trouble breathing) experienced by participants where score range is 0 (none) to 4 (very severe). BODE score is derived into a score range of 0 (healthy) to 10 (severe COPD).
Time Frame: Baseline and Week 53
Population: The mITT population included all participants who were randomized into the study and received any investigational product. Here, 'N' signifies those participants evaluable for this measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 123 | 116
units on a scale | -0.27 (0.107) | -0.08 (0.110)

7. Secondary Outcome: Percentage of Participants With Improvement in Body Mass Index, Airflow Obstruction, Dyspnea, and Exercise Capacity (BODE) Score
Description: The BODE index is a multi-dimension COPD grading system that incorporates body-mass index (B), degree of airflow obstruction (O), dyspnea (D), and exercise capacity (E) as measured by the modified medical research council (MMRC) dyspnea scale and the 6-minute walk test. The MMRC dyspnea scale is a 5-point scale that measures the level of dyspnea (trouble breathing) experienced by participants where score range is 0 (none) to 4 (very severe). BODE score is derived into a score range of 0 (healthy) to 10 (severe COPD). Negative change score signifies improvement compared to baseline. Number of participants with improvement in BODE score compared to baseline were reported.
Time Frame: Baseline and Week 53
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 123 | 116
percentage of participants | 39.0 | 33.6

8. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to Week 69 that were absent before treatment or that worsened relative to pre-treatment state. TEAEs reported below included both SAEs and non-serious AEs.
Time Frame: Day 1 up to Week 69
Population: Safety population included all participants who were randomized and received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 164 | 160
participants
  TEAEs | 130 | 130
  TESAEs | 35 | 41

9. Secondary Outcome: Observed Serum Concentrations of MEDI8968
Time Frame: Pre-dose (Baseline), Post-dose on Week 53
Population: PK population included all participants who were randomized, received at least one dose of investigational product, and had at least one post-dose serum concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliters (ng/mL)
Arm/Group | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 158
nanogram per milliliters (ng/mL)
  Baseline (n=145) | 1.7 (14.6)
  Week 53 (n=120) | 28555.7 (27545.6)

10. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies for MEDI8968 at Any Visit
Description: Anti-drug antibodies for MEDI8968 were analyzed for participants who received placebo or MEDI8968 as per planned analysis.
Time Frame: Day 1 up to Week 69
Population: Immunogenicity (IM) population included all participants who were randomized, received at least one dose of investigational product, and had at least one post-dose serum sample for IM testing.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI8968 600 mg IV, 300 mg SC
Number analyzed (Participants) | 163 | 157
participants | 10 | 19

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 69
Groups:
- MEDI8968 300 mg: MEDI8968 600 milligram (mg) as IV infusion on Day 1 followed by 300 mg injection SC every 4 weeks up to Week 5.
Arm/Group | PLACEBO | MEDI8968 300 mg
Serious Adverse Events (participants affected / at risk) | 35/164 | 41/160
Other Adverse Events (participants affected / at risk) | 127/164 | 122/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=164) | MEDI8968 300 mg (N=160)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Adams-stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ebstein's anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (29) | 18 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=164) | MEDI8968 300 mg (N=160)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 6 (6) | 8 (13)
Bronchitis (Infections and infestations) | 4 (4) | 5 (7)
Nasopharyngitis (Infections and infestations) | 11 (13) | 11 (12)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Sinusitis (Infections and infestations) | 5 (6) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (7) | 5 (8)
Weight decreased (Investigations) | 3 (3) | 4 (5)
Dyslipidaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 7 (27) | 10 (10)
Insomnia (Psychiatric disorders) | 5 (5) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 71 (138) | 64 (112)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 7 (10) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.